CLINICAL TRIAL: NCT05731713
Title: Discovering Our Story, to Develop the Journey of Transformation
Brief Title: Journey of Transformation Curriculum for Native American Youth
Acronym: JOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Teresa Evans-Campbell, Associate Professor: School of Social Work, University of Washington
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00012676-02; 1R01DA050521-01A1 (NIH)
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Drinking; Tobacco Use; Substance Use; Sexual Behavior
Keywords: Native American; American Indian; Adolescents
MeSH Terms: conditions — Alcohol Drinking; Tobacco Use; Substance-Related Disorders; Sexual Behavior

STUDY DESIGN:
Intervention Model Description: A stepped-wedge clinical trial with study participants recruited in staggered cohorts, with those in each annual recruitment wave receiving individual-level assignment to either immediate intervention or waitlist control.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate group (Experimental): Study participants in the immediate group will be randomly assigned to start the intervention immediately at the beginning of the fall trimester.
  Interventions: Behavioral: Journey of Transformation-Native Youth Health Leadership Program curriculum
- Waitlist group (Experimental): Study participants in the waitlist group will be randomly assigned to start the intervention at the beginning of the winter trimester.
  Interventions: Behavioral: Journey of Transformation-Native Youth Health Leadership Program curriculum

INTERVENTIONS:
Behavioral: Journey of Transformation-Native Youth Health Leadership Program curriculum — Curriculum activities will include traditional storytelling and other Native American cultural arts activities (i.e., drum making, film making), as well as Traditional Ecological Knowledge (TEK) activities and field trips. Curriculum content explains leadership skills and promotes healthy decision-making around substance use and sexual health.

SUMMARY:
The investigators will conduct a waitlist control trial to test the efficacy of the Journey of Transformation-Native Youth Health Leadership Program (JOT) in terms of delaying or reducing tobacco and other substance use and improving sexual health.

DETAILED DESCRIPTION:
This study assesses a new curriculum that will be available to students in the tenth grade. The lessons will include traditional storytelling and other Native American cultural arts activities (i.e., drum making, film making, field trips), as well as Traditional Ecological Knowledge (TEK) activities. This study also assesses how well the curriculum explains leadership skills, Native American cultural arts, the natural environment, and promotes healthy decision-making around health and relationships.

Participants are assigned to a health class that starts the curriculum in the fall or to a health class that will start the curriculum in the winter. Participants will:

Week 1. Complete a 15-20- minute online survey about healthy relationships, drug use, youth leadership skills, and connecting with Native communities.

Weeks 1 - 3. Meet with a study educator up to two times to set goals around health, healthy relationships and how to reduce or avoid alcohol, tobacco, or other drug use.

Weeks 1 - 12 (months 1-3). As part of the class, attend up to ten health sessions on healthy behaviors and health promotion. Learn new skills around youth leadership, storytelling, and traditional health practices. The sessions will highlight connection to tribal traditions.

Month 3. Complete an online check-in survey via a link sent to participants' email address.

Month 6. Complete an online check-in survey via a link sent to participants' email address.

Month 12. Complete an online check-in survey via a link sent to participants' email address.

Optional after school activities:

Weeks 9 - 16 (months 3-4). Attend a once-a-month activity to help build leadership skills. Activities are between 1-2 hours after school and include drum making, film making, creating a storytelling vest that incorporates their own cultural symbols, and up to two outdoor field trips. The field trips are to places of cultural significance near the school and involve a 30-45 minute hike.

Week 16 (month 4). Meet with the study educator for a session to revise goals for health and community leadership.

Weeks 9 - 24 (months 3-6). Attend a 2-hour digital storytelling training and three monthly planning sessions to prepare for an optional digital storytelling leadership night. Stories can be about what participants have learned about health promotion, traditional health practices, and to celebrate their health leadership journey.

Week 25 (month 6). Attend the leadership night and present digital stories if participants would like. Help prepare a traditional feast and giveaway that will honor community culture and values.

ELIGIBILITY:
Inclusion Criteria:

* Attends an off-reservation boarding school in the tenth grade at time of enrollment

Exclusion Criteria

* None

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 255 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in patterns of 30 day substance use assessed by self-report | Baseline to 3-month (post-intervention) follow-up; Baseline to 6-month follow-up; Baseline to 12-month follow-up (immediate group only)
  Patterns of substance use (Monitoring the Future [MTF] 30-day self-report assessed on an ordinal scale [0 occasions, 1-2 occasions, 3-5 occasions, 6-9 occasions, 10-19 occasions, 20-39 occasions, 40 or more occasions]). Substances include tobacco, alcohol, marijuana, stimulants, inhalants, opioids, and other drugs.
Change in sexual behavior assessed by self-report | Baseline to 3-month (post-intervention) follow-up; Baseline to 6-month follow-up; Baseline to 12-month follow-up (immediate group only)
  Primary sexual behaviors assessed by items from the Adolescent Sexual Activity Index

SECONDARY OUTCOMES:
Change in intentions to use alcohol, cigarettes, and marijuana in the next year (assessed by Monitoring the Future [MTF]) | Baseline to 3-month (post-intervention) follow-up; Baseline to 6-month follow-up; Baseline to 12-month follow-up (immediate group only)
  Assess intention to use alcohol, cigarettes, and marijuana in the next year (3 items) on a 5-point scale (I have already tried [substance], I definitely will, I probably will, I probably will not, I definitely will not). Scores are summed and standardized on a scale of 0 to 100 percent.
Change in the Specific Event Drug and Alcohol Refusal Self-Efficacy (SEDARE) Measure | Baseline to 3-month (post-intervention) follow-up; Baseline to 6-month follow-up; Baseline to 12-month follow-up (immediate group only)
  The Specific Event Drug and Alcohol Refusal Self-Efficacy (SEDARE) measure captures the perceived likelihood that youth will use drugs and alcohol in specific situations on a 3-point scale (Yes, No, Unsure). Higher scores reflect higher perceived ability to refuse alcohol or drugs.
Change in the Sexual Health and Reproductive Empowerment for Young Adults Scale (self-efficacy) (Upadhyay et al., 2020) | Baseline to 3-month (post-intervention) follow-up; Baseline to 6-month follow-up; Baseline to 12-month follow-up (immediate group only)
  23 items will be used to assess young people's empowerment regarding sexual and reproductive health on a 5-point Likert scale (Not at all true to Extremely true).

CONTACTS AND LOCATIONS:
Overall Officials: Teresa A Evans-Campbell, MSW, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified IPD will be available after institutional IRB and agency approval.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: De-identified data will be available for 12 months after publication of the main findings manuscript. Other resources, such as training materials and the curriculum, will be available after demonstration of their efficacy.
Access Criteria: Contact PI for access.

REFERENCES:
- [Background] Miech, Richard A., Johnston, Lloyd D., Bachman, Jerald G., O'Malley, Patrick M., Schulenberg, John E., and Patrick, Megan E. Monitoring the Future: A Continuing Study of American Youth (8th- and 10th-Grade Surveys), 2020. Inter-university Consortium for Political and Social Research [distributor], 2021-10-26. https://doi.org/10.3886/ICPSR38189.v1
- [Background] Belgrave FZ, Reed MC, Plybon LE, Corneille M. The impact of a culturally enhanced drug prevention program on drug and alcohol refusal efficacy among urban African American girls. J Drug Educ. 2004;34(3):267-79. doi: 10.2190/H40Y-D098-GCFA-EL74. PMID 15648887
- [Background] Upadhyay UD, Danza PY, Neilands TB, Gipson JD, Brindis CD, Hindin MJ, Foster DG, Dworkin SL. Development and Validation of the Sexual and Reproductive Empowerment Scale for Adolescents and Young Adults. J Adolesc Health. 2021 Jan;68(1):86-94. doi: 10.1016/j.jadohealth.2020.05.031. Epub 2020 Jul 17. PMID 32690468
- [Background] National Institute on Drug Abuse, University of Michigan, Institute for Social Research. (2016). Monitoring the Future, 2016 (Combined Forms - Part B). Ann Arbor, MI: Institute for Social Research, University of Michigan.